CLINICAL TRIAL: NCT00578370
Title: A Phase I, Single-Center, Randomized, Vehicle-Controlled Study, Double-Blind for the Study Preparations and Observer-Blind for the Comparators to Determine the Antipsoriatic Efficacy and Tolerability of Topical Formulations With Ciclosporin in a Psoriasis Plaque Test
Brief Title: Efficacy and Tolerability Study of Topical Ciclosporin in a Psoriasis Plaque Test
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ISDIN (Industry)
Responsible Party: ISDIN, ISDIN
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISD001-CI-07; 2007-002947-26
Record Dates: First submitted 2007-12-20; First posted 2007-12-21 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2008-11

CONDITIONS: Psoriasis
Keywords: Ciclosporin; Plaque type psoriasis; Psoriasis plaque test; Sonography; Cyclosporin; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Cyclosporine; Betamethasone; calcipotriene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: Ciclosporin 0.5% (Formulation 01B)
- 2 (Experimental)
  Interventions: Drug: Ciclosporin 1.5% (Formulation 02B)
- 3 (Active Comparator)
  Interventions: Drug: 0.1% betamethasone
- 4 (Active Comparator)
  Interventions: Drug: 0.005% calcipotriol
- 5 (Placebo Comparator)
  Interventions: Drug: Formulation 00B

INTERVENTIONS:
Drug: Ciclosporin 0.5% (Formulation 01B) — Cutaneous emulsion 200µl once a day (26 days)
  Arms: 1
Drug: Ciclosporin 1.5% (Formulation 02B) — Cutaneous emulsion 200µl once a day (26 days)
  Arms: 2
Drug: 0.1% betamethasone — Solution 200µl once a day (26 days)
  Other Names: Betnesol V crinale 0.1%
  Arms: 3
Drug: 0.005% calcipotriol — Solution 200µl once a day (26 days)
  Other Names: Daivonex solution 0.005%
  Arms: 4
Drug: Formulation 00B — Cutaneous emulsion (Vehicle to Formulation 01B and Formulation 02B) 200µl once a day (26 days)
  Arms: 5

SUMMARY:
Ciclosporin is a cyclic nonribosomal polypeptide of 11 amino acids produced by the fungi Tolypocladium inflatum and Cylindrocarpon lucidum. Ciclosporin is a highly efficient immunosuppressant drug widely used in post-allergenic organ transplant to reduce the activity of the subject's immune system and so the risk of organ rejection. Apart from transplant medicine, ciclosporin is also used in the treatment of autoimmune diseases like psoriasis and infrequently in rheumatoid arthritis and related diseases, although it is only used in severe cases.

Ciclosporin blocks the lymphocytes, especially the T-lymphocytes, in the G0- or G1-phase of the cell cycle. Moreover it inhibits the production and release of lymphokines including interleukin 2 or the T-cell growth factor.

Generally ciclosporin is taken orally (capsule or solution)or by injection in doses of 1.5 to 5.5 mg/kg/day. In the topical cutaneous emulsion presented here, ciclosporin is available at a concentration of 0.5 and 1.5%.

The purpose of this study is the demonstration of antipsoriatic efficacy and tolerability of topical cutaneous ciclosporin in subjects with psoriasis vulgaris.

DETAILED DESCRIPTION:
Psoriasis is a common dermatological disorder, consisting of both an inflammatory and a hyperproliferative component. Scaly, erythematous infiltrated skin lesions are indicative of psoriasis vulgaris. The disease is characterized micromorphologically by epidermal hyperplasia with incomplete differentiation, intraepidermal accumulation of polymorphonuclear neutrophils, elongated papillae containing dilated, tortuous capillaries and lymphohistiocytic infiltrate.

Since the underlying cause of the disease remains unknown, causal therapy is not possible. The complex clinical picture necessitates a polypragmatic therapeutic approach. Typical therapies include phototherapy and photochemotherapy, topical treatment with corticosteroids, vitamin D3 analogs, coal-tar preparations and dithranol, and systemic treatment with retinoids, methotrexate and ciclosporin (oral or injection).

In the present study the topical cutaneous ciclosporin formulation for topical treatment of psoriasis will be tested in low-dose for efficacy and tolerability. Two concentrations of the ciclosporin formulation (0.5% and 1.5%), the corresponding vehicle, a marketed corticoid preparation and a marketed topical Vitamin-D-analog will be tested simultaneously in the same patient. Five test fields located at the torso and at the extremities will be examined per subject, and will be treated non-occlusively on 22 study days over a period study of 26 days.

Experimental measurements (sonography) and clinical assessments will be performed at baseline and on some study days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic plaque type psoriasis
* Sexually active females of childbearing potential should either be surgically sterile (hysterectomy or tubal ligation), or should use a highly effective medically accepted contraceptive regimen

Exclusion Criteria:

* Local treatment with antipsoriatics (except for salicylic acid in vaseline) in the 4 weeks preceding and during the study (corticosteroids 8 weeks)
* Systemic treatment with antipsoriatics or therapy with PUVA, selected ultraviolet photo therapy in the three months preceding and during the study
* Treatment with systemic or locally acting medications which might counter or influence the study aim
* Previous therapy with methotrexate over many years
* Therapy with nephrotoxic medication
* Therapy with digoxin, colchicin and statins
* Medications which might influence the potassium metabolism
* Subjects with known dysfunction of the calcium metabolism
* Subjects with increased uric acid or potassium serum levels
* Erythrodermic psoriasis, psoriasis punctata and pustular psoriasis or extended chronic stationary forms of psoriasis
* Subjects with acute virus infection
* Subjects with acne, anogenital pruritus, rosacea, perioral dermatitis, specific skin problems (skin tuberculosis, luetic skin diseases), vaccination reactions, skin infections caused by bacteria or viruses
* Symptoms of a clinically significant illness that may influence the outcome of the study in the four weeks before and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Psoriatic infiltrate measured by sonography | 26 days

SECONDARY OUTCOMES:
Skin condition measured by scoring | 26 days

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Gassmueller, MD, Principal Investigator — Bioskin GmbH
Locations (1):
- Bioskin, Hamburg, Hamburg, Germany

REFERENCES:
- [Background] Dumas KJ, Scholtz JR. The psoriasis bio-assay for topical corticosteroid activity. Acta Derm Venereol. 1972;52(1):43-8. No abstract available. PMID 4111105
- [Background] Wendt H, Frosch PJ. Psoriasis-Plaque Test. 31 - 35 in: Clinico-pharmacological models for the assay of topical corticoids. Wendt H, Frosch PJ (eds.) 1982, Karger Verlag, Basel